CLINICAL TRIAL: NCT00549952
Title: Observational Study of Anti-Cancer Therapy Induced Oral Mucositis in Korean Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 256-KOB-0701
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention study

SUMMARY:
to survey oral mucositis after chemotherapy and Concurrent chemoradiotherapy in Korean cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with one cancer among head and neck cancer, esophageal cancer, breast cancer, colorectal cancer, gastric cancer, and non-small cell lung cancer, who are being treated or going to be treated as one between A and B A. Chemotherapy only B. Concurrent chemoradiotherapy

Exclusion Criteria:

* Patients who are pregnant or breast feeding, absent from effective(medically proven) contraceptive method for females of childbearing potential
* Patients with performance status of ECOG score is more than 3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
incidence and severity of oral mucositis

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University hospital, Seoul, South Korea